CLINICAL TRIAL: NCT00715000
Title: Prevention of Dehydration in Premature Babies Between 32 and 34+6 Gestational Age, Weighing Between 1700 and 2200 g, During the First Days of Life, Using Oral Rehydration Solution in Alternative to Intravenous Infusion
Brief Title: Oral Versus Intravenous Rehydration for Prevention of Dehydration in Premature Babies, During the First Days of Life.
Acronym: SROPREMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060208
Record Dates: First submitted 2008-07-11; First posted 2008-07-14 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Low Birth Weight Infant; Enteral Nutrition
Keywords: Preterm babies hydration; Oral rehydration solution; Continuous gastric drip; Fluid therapy; Premature babies comfort; Infant care; Technical challenge for the nurses/doctors in charge
MeSH Terms: conditions — Osteoarthritis | interventions — Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): SRO
  Interventions: Procedure: Oral rehydration therapy
- 2 (Active Comparator): classical hydration via intravenous infusion
  Interventions: Procedure: classical hydration via intravenous infusion

INTERVENTIONS:
Procedure: Oral rehydration therapy — oral rehydration solution
  Other Names: SRO
  Arms: 1
Procedure: classical hydration via intravenous infusion — intravenous infusion
  Other Names: IV
  Arms: 2

SUMMARY:
This prospective randomised study comparing administration of a hypo-osmolar oral hydration solution with the classical hydration via IV (intravenous) infusion in premature infants of more than 32 weeks GA (gestational age) aims to determine whether administration of a hypo-osmolar oral hydration solution is as efficient as intravenous infusion.

DETAILED DESCRIPTION:
In order to prevent dehydration of the premature infant during the first days of life, enteral nutrition with milk must be complemented by an additional fluid supply, commonly administered intravenously. We propose to perform a prospective randomised multi-centric study comparing administration of a hypo-osmolar oral hydration solution with the classical hydration via IV (intravenous) infusion in premature infants of more than 30 weeks GA (gestational age).

We define success as a weight loss inferior to 15 % of birth weight and a weight at day 15 superior to birth weight. Failure was defined hence as a weight loss superior to 15% of birth weight or a weight at day 15 inferior to birth weight or a severe complication or death. Major violations of the protocol in the study group will be counted as failures. The other objectives were to determine whether oral hydration demonstrates practical advantages: less complications in initial management, more comfort for the baby and less technical challenges for the nurses/doctors in charge. Furthermore to evaluate the clinical tolerance of oral hydration from a nutritional point of view and to examine it's effects on intestinal function (defecation, gastric residues), signs of intestinal inflammation and GI flora.

ELIGIBILITY:
Inclusion Criteria:

* Premature babies between 32 to 34 + 6 weeks of gestation, with a birth weight greater than 1700g and less than 2200g under exclusion of SGA (small for gestational age) babies with a BW < 10th percentile.
* Infants must be included within the first 12 to 24 hours of life
* Good tolerance to nasogastric milk feeding
* Necessity of additional fluid supply
* Any suspicion of gastro intestinal or metabolic disease
* Maximal humidity in incubator
* Parental consent form

Exclusion Criteria:

* suspicion of gastro-intestinal disease,
* severe digestive risks, and metabolic diseases in the family history,
* metabolic or hydro-electrolyte disorders
* other severe diseases

Ages: 32 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2008-07; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Weight | Day 0 to day 16 or day of recovering original birth day

SECONDARY OUTCOMES:
Weight, length, head circumference and brachial circumference | day 3, 15 of life, and at 37 GA.
Weight, Height/length, head circumference and brachial circumference | 6 and 12 months
pathologic digestive diseases (enteropathy, NEC…) | J0 to J16
metabolic tolerance during the first week of life: - hypoglycemia - fructose intolerance - bilirubin, electrolytes and creatinin level in blood | during the first week of life
pain and discomfort score (EDIN) evaluated 3 times a day | Day 0 to day 16
secondary IV infusion effects | Day 0 to day 8
number of failure to pick and to perfuse a baby | Day 0 to day 8
ORS culture | in case of infection
Adverse Events | Up to 12 months
Intestinal motility: - gastric residue - first meconium - first normal stool - number of stools during the first days of life | the first two weeks of life

CONTACTS AND LOCATIONS:
Overall Officials: Hasini RAZAFIMAHEFA, MD, Principal Investigator — Assistance Publique-Hôpitaux de Paris, Hôpital Antoine Béclère
Locations (1):
- Assistance Publique - Hôpitaux de Paris Hôpital Antoine Béclère, Clamart, France